CLINICAL TRIAL: NCT01062308
Title: The Effectiveness of Taping Technique Versus Conventional Techniques in Prevention of Shoulder Injuries in Patients With Acute Stroke-A Prospective, Randomized, Interventional, Outcome Blinded (PROBE Design), Parallel Design Trial
Brief Title: STRIPS: Shoulder Taping Reduces Injury and Pain in Stroke
Acronym: STRIPS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Christian Medical College and Hospital, Ludhiana, India (Other)
Collaborators: Uppal Neuro Hospital (Other); Heart and Brain Center, Guntur, Andhra Pradesh, India (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Jeyaraj Pandian; CMC/NEU/COP/JDP/2009/001 (Other: CMC Ludhiana)
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Results first posted 2013-03-07 (Estimated); Last update posted 2013-03-12 (Estimated); Status verified 2013-03

CONDITIONS: Stroke; Shoulder Injury
Keywords: Stroke; Taping; Pain; Shoulder Injury
MeSH Terms: conditions — Stroke; Shoulder Injuries; Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Taping (Experimental): The tri-pull method of taping was used.Taping was initiated by first applying three, two-inch wide and approximately ten-inch long, pieces of elastic adhesive tape strips. The first strip was applied from the mid-humerus deltoid tuberosity across the scapula. The second strip was applied from the deltoid tuberosity across the clavicle to the mid-clavicle, but before the supra-sternal notch. The third strip was placed from the deltoid tuberosity over the acromion process to the neck.
  Interventions: Procedure: Taping and Sham Taping
- Sham Taping (Active Comparator): This was done using the same tapes. Three strips of tapes were applied in same position without repositioning the joint. All other Physiotherapy measures like positioning, handling technique and range of motion exercises were equally done for both the groups.
  Interventions: Procedure: Sham Taping

INTERVENTIONS:
Procedure: Taping and Sham Taping — Taping shoulder with Hospiplast tape.
  Taping the shoulder after acute stroke to prevent shoulder injury and pain.
  Taping the shoulder after acute stroke and compare with sham taping group.
  Treatments:
  1. Positioning technique
  2. Handling technique
  3. Range of motion exercises
  4. Taping technique
  Other Names: Shoulder Taping in Stroke
  Arms: Taping
Procedure: Sham Taping — Shoulder Taping for 14 days which will be changed after every 3 days.
  Arms: Sham Taping

SUMMARY:
Background and Rationale: The most commonly seen disabilities in stroke patients are shoulder injuries such as shoulder pain, glenohumeral subluxation, spasticity of shoulder muscles, soft-tissue trauma, rotator cuff tears, and shoulder-hand syndrome.

Taping is widely used in the field of rehabilitation as both means of treatment and prevention of sports related injuries. Scarce information is available regarding the use of shoulder taping in preventing shoulder injuries in stroke patients. Aims:

To find out the effectiveness of taping technique with conventional treatment versus sham taping and conventional treatment in prevention of shoulder injuries in patients with acute stroke.

Hypothesis:

Taping technique with conventional treatment will be superior to conventional treatment alone in preventing shoulder injuries in patients with acute stroke.

Methods Research setting: Stroke unit, department of Neurology, Christian Medical College (CMC) Ludhiana, Punjab, India and College of Physiotherapy, CMC Ludhiana.

Study design: prospective, randomized, outcome blinded trial (PROBE design). Study period: Prospective for 18 months from May 2009 All stroke patients with upper limb weakness within 48 hours after the ictus and with Brunnstrom's stage of recovery 1 and 2 will be included in the study. Patients will be randomized into two groups using lottery method. The treatment arm group(Group I) include shoulder taping with conventional techniques that is(positioning, handling technique and passive range of motion exercises) and the control arm (Group II) include sham taping with conventional techniques with sham taping. A total of 80 patients in each group will be included. The plastic micropore and elastic adhesive tape will be used for taping the affected shoulder. The sham taping will be done using the same tapes but without stretching the concerned muscles and joints. The tapes will be changed every 3 days and will remain for 14 days. The outcome measures are as follows; Primary: Pain: Visual Analog Scale and Activities of daily living: Shoulder Pain and Disability Index (SPADI); Secondary: Range of motion: using a Goniometer. The outcome will be assessed by an independent physiotherapist who will be blinded to the clinical details. Patients will be followed-up at 14 days and 30 days. Statistical analyses will be done using SPSS software version 16.

DETAILED DESCRIPTION:
Background and Rationale:

Stroke is the second leading cause of death and a major cause of disability worldwide. Two-thirds of stroke deaths worldwide occur in developing countries. According to recent reports from India the incidence and 30-day case fatality rates are higher than the developed countries. In both rural and urban India there has been a rise in the non-communicable diseases like stroke and coronary artery disease. In developing countries the average age of stroke is 15 years less than that of developed countries.

It has been estimated that by 2021, the stroke related "disability adjusted life years" (DALY) would become 61 million, and 52 million would be in developing nations. According to recent studies 55-70% of stroke survivors become fully independent by one year and 7-16% remain completely disabled. Prominent residual spasticity occurs in 46% of patients.

Shoulder Injuries in Stroke The most commonly seen disabilities in stroke patients are shoulder injuries which are more common during sub-acute phase of stroke. Pain in the affected shoulder often referred to as hemiplegic shoulder pain, is a common complication. The other types of shoulder injuries include glenohumeral subluxation, spasticity of shoulder muscles, soft-tissue trauma, rotator cuff tears, and shoulder-hand syndrome or reflex sympathetic dystrophy. Shoulder injuries can negatively affect rehabilitation outcomes as good shoulder function is a pre-requisite for successful transfers, maintaining balance, performing activities of daily living and for effective hand function.

Biomechanics of shoulder injuries in stroke patients A stroke patient with upper limb weakness tends to place the arm in a resting position and this promotes shortening of the shoulder adductors and internal rotators, and the elbow, wrist and hand flexors. This habitual posturing of the upper limb can result in adaptive changes to muscle tissue that impede both passive and active joint movement.As motor power returns, the pattern of recovery may be imbalanced, with individual muscles developing strength at different rates or there may be increased tone in certain muscle groups. Imbalanced motor return and persistent attempts to move with increased activation of just one muscle group can pull the scapula and humerus into abnormal postures. When this posture is maintained, the resting length of the surrounding muscles may either shorten or lengthen, thereby disrupting the normal biomechanics of that joint. In addition in flaccid stage, the scapula assumes a depressed and downward rotated position, as the paretic serratus anterior and upper part of trapezius muscle no longer support the scapula. The combination of flaccid supportive musculature and a downward rotated scapula predisposes the head of humerus to undergo inferior subluxation relative to the glenoid fossa.

Treatment options for shoulder injuries in stroke patients The ideal management of hemiplegic shoulder pain is to prevent it happening in the first place. Various strategies have been employed in the prophylaxis of hemiplegic shoulder pain. For prophylaxis to be effective, it must be begin immediately after the stroke. Early passive shoulder range of motion, and supporting and protecting the involved shoulder in the early flaccid stage, local treatments such as heat and cold therapy, transcutaneous electrical nerve stimulation, functional electrical stimulation, range of motion exercises, EMG biofeedback are regarded as important steps to reduce the development of shoulder pain. Careful positioning and handling of the limb are thought to prevent hemiplegic shoulder pain, but there is a range of opinions about how correct limb positioning is best achieved. Careful positioning of the shoulder serves to minimize subluxation and later contractures as well as possibly promote recovery, while poor positioning may adversely affect symmetry, balance and body image. Through correct positioning, the development of shoulder pain can be prevented. However, the effectiveness of any of these methods in preventing shoulder injuries has yet to be established.

Taping is widely used in the field of rehabilitation as both means of treatment and prevention of sports related injuries.The essential function of tape is to provide support during movement. Taping is a treatment method used in conjunction with other therapeutic techniques in the treatment of various musculoskeletal and neuromuscular deficits. It helps to support or inhibit muscle function, support joint structure, reduce soft tissue inflammation, and reduce pain. It also can produce feedback to the muscle to maintain preferred postural alignment. Various taping materials have been used in rehabilitation (Kinesio tape, Leukotape, Cover-roll stretch tape).

Scarce information is available regarding the use of shoulder taping in preventing shoulder injuries in stroke patients. Peters and Lee, 2003 studied a single stroke patient during the sub-acute phase of stroke. The patient reported decrease in pain, improvement in activities of daily living and range of motion of the shoulder. However there are no controlled studies using large number of stroke patients. Moreover the effectiveness of taping in conjunction with other therapeutic activities to facilitate improvement in restoring functional use of the upper extremity during the acute phase of stroke has not been studied. Shoulder taping may prove to be economically sensible by preventing shoulder subluxation which would decrease the number of therapy treatment sessions. Taping materials are locally available and it could be an affordable solution to prevent shoulder injuries following stroke.

Study goal, objectives and main research questions:

To find out the effectiveness of shoulder taping technique with conventional treatment versus sham taping and conventional treatment in prevention of shoulder injuries in patients with acute stroke.

Methods

Setting:

Stroke Unit, Department of Neurology, and College of Physiotherapy, Christian Medical College and Hospital, Ludhiana

Study design: Prospective, randomized, outcome blinded trial (PROBE design).

Sample size and sampling techniques:

A target sample size of 160 was chosen to provide 90% power (alpha=0•.05) with 25% drop-out to detect a minimum reduction in VAS of 38 in the intervention group based on the assumption that mean reduction in VAS score is 27 (SD 18) in control group. The sample size of 160 also had 90% power (alpha=0•.05) with 25% drop-out to detect a minimum of 20 reduction in SPADI score in the intervention group based on the assumption that mean reduction in SPADI score is 12 (SD12) in control group.

All consecutive stroke patients who give consent will be randomised in a blinded fashion to two treatment groups using lottery method. .

Patient groups The randomization will be done by an office personnel who will be unaware of the clinical details of the patients Group 1: patients will be given conventional treatment i.e. positioning, handling technique, passive range of motion exercises and taping of the affected shoulder Group 2: patients will be given conventional treatment alone which includes sham taping of the affected shoulder

Study definitions Stroke will be defined as per WHO: Syndrome of rapidly developing symptoms and signs of focal, and at times global, loss of cerebral function lasting more than 24 hours or leading to death, with no apparent cause other than that of vascular origin.

All stroke patients within first 48 hours after the onset of symptoms will be approached for inclusion

Instruments/tools Pain: Visual Analog Scale Range of motion: full circle universal Goniometer Activities of daily living: Shoulder Pain and Disability Index Stroke severity: National Institute for Health Stroke Scale34 Taping: Plastic micropore and elastic adhesive tape (Leucoplast) Brunnstrom stage of stroke recovery Glasgow coma scale

Techniques/ methods

Treatments

1. Positioning technique
2. Handling technique
3. Range of motion exercises
4. Taping technique Primary Outcome

1. VAS 2. SPADI

Secondary outcome:

ROM

Data management and analysis plan:

Data entry operator will enter the patient data. Statistical Analyses will be done using SPSS software version 16. Summary statistics including frequency, mean and standard deviation of variables of interest will be generated. Comparison of means of the continuous variables between the two treatment groups will be done using Student-t test, and the binary variables using Chi-square test. The means of the outcome measures (scores of visual analog scale, range of movements of shoulder and shoulder pain and disability index) at admission will be compared with the values at day 14 and day 30 using Student-t test between the two groups. A p value of <0.05 will be considered significant.

Implications of study results on patient safety practice and/or interventions

This study will be using locally available tapes such as plastic micropore and elastic adhesive tapes for taping the shoulder. They are easily available.

The results of this study has wider application if the taping technique is found effective, particularly in developing countries where resources are sparse. This simple technique will prevent stroke disability due to shoulder injuries and help in rehabilitation of stroke victims.

ELIGIBILITY:
Inclusion Criteria:

1. Stroke patients both ischemic and hemorrhagic with upper limb weakness within 48 hours after the ictus
2. Age over 18 years
3. Brunnstrom's stage of recovery 1 and 2
4. Patients willing to participate in the study

Exclusion Criteria:

1. Patients with Glasgow coma scale of <7
2. Patients on ventilator
3. Uncooperative patients
4. Patients having previous history of shoulder injury
5. Patients with Wernicke's aphasia
6. Patients having previous history of shoulder pain
7. Any previous history of skin allergy to tape

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2009-08; Primary Completion 2012-03 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeyaraj D Pandian, MD DM FRACP, Principal Investigator — Christian Medical College, Ludhiana
Locations (2):
- India (2):
  - Christian Medical College, Ludhiana, Punjab
  - Jeyaraj D Pandian, Ludhiana, Punjab

REFERENCES:
- [Derived] Pandian JD, Kaur P, Arora R, Vishwambaran DK, Toor G, Mathangi S, Vijaya P, Uppal A, Kaur T, Arima H. Shoulder taping reduces injury and pain in stroke patients: randomized controlled trial. Neurology. 2013 Feb 5;80(6):528-32. doi: 10.1212/WNL.0b013e318281550e. Epub 2013 Jan 23. PMID 23345636

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first Recruitment: Sep.2009 Date of Completion: March 2012
Groups:
- Taping: Procedure for preventing shoulder injury
- Sham Taping: Sham Taping was applied without stretching the concerned muscles.
Period: Overall Study
Arm/Group | Taping | Sham Taping
Started | 80 | 82
Completed | 64 | 72
Not Completed | 16 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Taping | Sham Taping | Total
Number analyzed (Participants) | 80 | 82 | 162
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 64 | 59 | 123
  >=65 years | 16 | 23 | 39
Age Continuous [Mean (Standard Deviation); unit: years] | 56 (13) | 60 (13) | 58 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 33 | 56
  Male | 57 | 49 | 106
Region of Enrollment [Number; unit: participants]
  India | 80 | 82 | 162

OUTCOME MEASURES:

1. Primary Outcome: Pain: Visual Analog Scale
Description: Visual analog scale (VAS) is an 11-point scale displayed on a 100 mm horizontal line, ranging from 0 ("No Pain") to 100 ("Worst Pain Imaginable") Shoulder pain and disability index (SPADI) is a 13-item questionnaire that consists of 2 subscales for pain (5 items) and disability (8 items), which is scored by taking an average of the 2 subscales. Scores range from 0 to 100, with higher scores indicating greater pain and disability
Time Frame: 14 days and 30 days
Population: On the basis of complete follow up
Measure: Mean (95% Confidence Interval); unit: mm
Arm/Group | Taping | Sham Taping
Number analyzed (Participants) | 65 | 72
mm
  VAS Baseline to day 14 | -2.3 [-9.3 to 4.7] | 1.4 [-5.3 to 8]
  VAS baseline to day 30 | -9.2 [-17 to -1.4] | 2.6 [-4.8 to 10.1]
Statistical Analysis 1: Comparison: Taping vs Sham Taping; Test type: Superiority or Other; p = 0.03, Mixed Models Analysis; Mean difference from baseline to day 30 = -11.8, 95% CI 2-sided [-22.6 to -1.1]

2. Secondary Outcome: Passive Range of Motion (ROM)
Description: Passive range of motion (ROM) of shoulder was measured with full circle goniometer. The normal range of movement of flexion and abduction is 180 degree.
Time Frame: 14 days and 30 days
Population: On the basis of follow up completion
Measure: Mean (95% Confidence Interval); unit: degree
Arm/Group | Taping | Sham Taping
Number analyzed (Participants) | 64 | 72
degree
  ROM baseline to day 14 | 2.9 [-3.5 to 9.4] | -4.1 [-10.2 to 2]
  ROM baseline to day 30 | 4.9 [-1.8 to 11.7] | -1.7 [-8.1 to 4.7]
Statistical Analysis 1: Comparison: Taping vs Sham Taping; Test type: Superiority or Other; p = 0.16, Mixed Models Analysis; Mean difference from baseline to day 30 = 6.6, 95% CI 2-sided [-2.7 to 15.9]

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Taping | Sham Taping
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/72
Other Adverse Events (participants affected / at risk) | 0/65 | 0/72

LIMITATIONS AND CAVEATS:
Follow up period was short. Secondly, X rays of the shoulder were not done to document other shoulder injuries.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No